CLINICAL TRIAL: NCT06749093
Title: Health Effects of Wood Smoke and Traffic-Related Air Pollution Exposures: a Necessary Comparison
Acronym: WADE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Christopher Carlsten, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: H24-00776
Record Dates: First submitted 2024-10-23; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Healthy Individuals; Allergic Rhinitis
Keywords: Air Pollution; Wood Smoke; Diesel Exhaust
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Vehicle Emissions; Air Pollution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Filtered Air (FA) (Placebo Comparator): Participants will be exposed to 2 hours of high-efficiency particulate air (HEPA) filtered air (FA).
  Interventions: Other: Filtered Air (FA)
- Wood Smoke (WS) (Active Comparator): Participants will be exposed to 2 hours of controlled wood smoke (WS) standardized to 300ug/m^3 of particulate matter with a diameter of 2.5 micrometers or less (PM2.5).
  Interventions: Other: Wood Smoke (WS)
- Diesel Exhaust (DE) (Active Comparator): Participants will be exposed to 2 hours of controlled diesel exhaust (DE) as a model of traffic-related air pollution (TRAP) standardized to 300ug/m^3 of particulate matter with a diameter of 2.5 micrometers or less (PM2.5).
  Interventions: Other: Diesel Exhaust (DE)
- Diesel Exhaust and Wood Smoke (DEWS) (Active Comparator): Participants will be exposed to 2 hours of combined controlled diesel exhaust (DE) and wood smoke (DEWS) standardized to 300ug/m^3 of particulate matter with a diameter of 2.5 micrometers or less (PM2.5).
  Interventions: Other: Diesel Exhaust and Wood Smoke (DEWS)

INTERVENTIONS:
Other: Filtered Air (FA) — Exposure to HEPA filtered air, as a control
  Arms: Filtered Air (FA)
Other: Wood Smoke (WS) — Wood smoke (WS) standardized to 300µg/m³ of particulate matter with a diameter of 2.5 micrometers or less (PM2.5).
  Arms: Wood Smoke (WS)
Other: Diesel Exhaust (DE) — Diesel exhaust (DE) standardized to 300µg/m³ of particulate matter with a diameter of 2.5 micrometers or less (PM2.5).
  Other Names: Traffic-Related Air Pollution
  Arms: Diesel Exhaust (DE)
Other: Diesel Exhaust and Wood Smoke (DEWS) — Combined diesel exhaust and wood smoke standardized to 300µg/m³ of particulate matter with a diameter of 2.5 micrometers or less (PM2.5).
  Other Names: Air Pollution
  Arms: Diesel Exhaust and Wood Smoke (DEWS)

SUMMARY:
Accumulating evidence demonstrates that breathing air pollutants leads to devastating increases in sickness and death worldwide over time. However, there is little data comparing the effects of different types of air pollution on health. In Canada, traffic-related air pollution and wood smoke (wildfires and wood burning for heating) are very common air pollutants. This study aims to safely complete a controlled human exposure study to test how these air pollution types acutely affect health.

DETAILED DESCRIPTION:
Healthy adult participants (total 48; 24 of each biological sex assigned at birth) will breathe filtered air (control), wood smoke (WS), diesel exhaust (DE), and DE plus WS (DEWS) each for 2 hours, with 4 weeks between each exposure (washout). Before and after each exposure, participants will answer questions, perform breathing tests, and give blood samples. At 24 hours after each exposure, participants will undergo a bronchoscopy to collect samples from their lungs.

The study will look at what (if any) are the differences between breathing in fresh air (filtered air - FA) or polluted air containing either wood smoke (WS), diesel exhaust (DE) or diesel exhaust plus wood smoke (DEWS). The research team will use wood smoke generated from pine wood, since it is one of the most common types of wood found in Western Canadian forests where forest fires occur.

The investigators will evaluate multiple endpoints as detailed in the Outcome Measures section. For each applicable endpoint, the investigators will evaluate stratified analyses and effect modification by biological sex, participant age, gene score, and microbiomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-40
* Healthy, with no history of respiratory disease
* Lifetime non-smoker and non-vaper.

Exclusion Criteria:

* Pregnant, planning to become pregnant, or breastfeeding during the study period (confirmed through pregnancy tests at each visit if applicable)
* Frequent WS or DE exposures (e.g. home fireplace used for heating/cooking, or employment in transportation, mining, or as a firefighter).

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Woodsmoke (WS) and/or diesel exhaust (DE) exposure effects on inflammatory cells in the lungs. | Comparison of the different arms (over the span of ~5 months).
  Differentially count lung cells.
Within-individual change in lung transcriptomic biomarkers of inflammation following exposure to woodsmoke and/or diesel exhaust. | Through study completion, anticipated ~5 months.
  Within-individual change in lung biomarkers of inflammation (serum amyloid A (SAA), c-reactive protein (CRP), chemokine ligand 18 (CCL18), and fibrinogen) in RNA.
Within-individual change in lung protein biomarkers of inflammation following exposure to woodsmoke and/or diesel exhaust. | Through study completion, anticipated ~5 months.
  Within-individual change in lung biomarkers of inflammation (serum amyloid A (SAA), c-reactive protein (CRP), chemokine ligand 18 (CCL18), and fibrinogen) in protein.
Within-individual change in circulating transcriptomic biomarkers of inflammation following exposure to woodsmoke and/or diesel exhaust. | Through study completion, anticipated ~5 months.
  Within-individual change in circulating biomarkers of inflammation (CX3CL1, CCL23, CXCL8, SAA, MMP9, MMP12, APOB, APOM, SOD1, NQO1, HMOX1, CAT, CYP1B1, CYP1A2, NFE2L2 and AHRR) in RNA.
Within-individual change in circulating protein biomarkers of inflammation following exposure to woodsmoke and/or diesel exhaust. | Through study completion, anticipated ~5 months.
  Within-individual change in circulating protein biomarkers of inflammation (CX3CL1, CCL23, CXCL8, SAA, MMP9, MMP12, APOB, APOM, SOD1, NQO1, HMOX1, CAT, CYP1B1, CYP1A2, NFE2L2 and AHRR).
Within-individual change in airway resistance following exposures to woodsmoke and/or diesel exhaust. | Through study completion, anticipated ~5 months.
  Within-individual change in airway resistance, as measured by impulse oscillometry (resonant frequency (Fres) and peripheral airway resistance (R5-R20)) across exposures to woodsmoke and/or diesel exhaust relative to filtered air.

SECONDARY OUTCOMES:
Woodsmoke (WS) and/or diesel exhaust (DE) exposure effects on inflammatory cells in the nose. | Comparison of the different arms (over the span of ~5 months).
  Differentially count nasal cells.
Within-individual changes in exhaled nitric oxide following woodsmoke (WS) and/or diesel exhaust (DE) exposures. | Comparison of the different arms (over the span of ~5 months).
  Measurement of fractional exhaled nitric oxide (FeNO) in parts per billion (ppb).
Woodsmoke (WS) and/or diesel exhaust (DE) exposure effects on symptoms, stress and perceptions. | Comparison of the different arms (over the span of ~5 months).
  Visual analog score (0-100) questionnaire will be completed, with a higher score indicating a worse outcome.
Woodsmoke (WS) and/or diesel exhaust (DE) exposure effects on lung function. | Comparison of the different arms (over the span of ~5 months).
  Lung function as evaluated by spirometry (e.g. FEV1).
Woodsmoke (WS) and/or diesel exhaust (DE) exposure effects on nasal resistance. | Comparison of the different arms (over the span of ~5 months).
  Measurement of peak nasal inspiratory flow (PNIF).

CONTACTS AND LOCATIONS:
Overall Officials: Chris Carlsten, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Participant data that underlie the results reported in accepted articles for publications, after deidentification (text, tables, figures, and appendices).
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal to the PI to complement the approved study aims.